CLINICAL TRIAL: NCT02945865
Title: Systematic Pain Assessment in Nursing Home Residents With Advanced Dementia; Effect on Pain Management and Patient Outcomes
Brief Title: Systematic Pain Assessment in Nursing Home Residents With Advanced Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Liv Halvorsrud, Associate Professor, PhD, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK 2014/1431
Record Dates: First submitted 2016-10-12; First posted 2016-10-26 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Pain; Dementia; Quality of Life
MeSH Terms: conditions — Pain; Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ITreatment arm: Pain Assessment (Experimental): Pain assessment by Doloplus-2 pain scale regularly and additional pain assessment in situations where pain is suspected.
  Interventions: Other: Pain assessment
- Control arm: No treatment (No Intervention): Treatment us usual

INTERVENTIONS:
Other: Pain assessment — Pain assessment with assessment tools
  Arms: ITreatment arm: Pain Assessment

SUMMARY:
It is estimated that 45-80 % of nursing home residents have substantial pain at any given time. Residents with impaired cognition have been found to report chronic pain more often, more frequent and more severe, compared to residents with normal cognition. Approximately 3/4 of permanent residents in nursing homes in Norway have developed dementia. The burden of dementia is often compounded by painful conditions. Despite over a decade of research on the subject, inadequate pain assessment and management remain significant problems among institutionalized older adults, with and without dementia. The poor pain management in patients with dementia has been attributed, at least in part, to difficulties with, and lack of, pain assessment in this population. Therefore, this study seek to determine the effect of regular pain assessment.

DETAILED DESCRIPTION:
The aim of the study is to determine the effect of regular pain assessment on pain management interventions applied and patient outcomes among patient with severe dementia.

A cluster randomized controlled trial will be conducted. A cluster is defined as a single independent nursing home. The clusters will be randomly assigned to either the experimental or control condition. Appropriate information will be given to both the intervention and the control group. All nurses in the experimental conditions will be taught how to administer the DOLOPLUS-2. The study will start after the initial education session. During the 3-month study period, the participating nursing staff will be asked to complete the DOLOPLUS-2 regularly. The control groups will receive standard methods of care. Data collection at baseline and at 4, 8 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years old
* Dementia diagnosis
* Severe language impairment/non-communicative
* Clinically significant pain and/or behavioral symptoms: a score of at least 44 on the Norwegian version of the Cohen-Mansfield Agitation Inventory (CMAI),
* or a score of at least 4 (frequency × severity) on items of the Neuropsychiatric Inventory - Nursing Home Version (NPI-NH),
* or an indication of clinically significant pain (≥ 5) according to the DOLOPLUS-2 at baseline

Exclusion Criteria:

* Short term stay, < 4 weeks
* Primary psychiatric diagnosis
* Delirium

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-01-26 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2018-03-17 (Actual)

PRIMARY OUTCOMES:
Change in analgesic intake measured in Defined Daily Dose (DDD) or a similar measure from baseline to 12 weeks. Will be assessed in both the Intervention and Control group. | 12 weeks
Change in pain score on the Dolplus-2 pain scale, and change in proportion scoring ≥ 5 on the Doloplus-2 scale from baseline to 12 week. Will be assessed in both the Intervention and Control group. | 12 weeks

SECONDARY OUTCOMES:
Change in psychotropic drug use from baseline to 12 weeks. Will be assessed in both the Intervention and Control group | 12 weeks
Change in NPS from baseline to 4, 8, 12 weeks. Will be assessed in both the Intervention and Control group | 4, 8, 12 weeks
Change in agitation measured with Brief Agitation Rating Scale (BARS) from baseline to 4 to 8 to 12 weeks. Will be assessed in both the Intervention and Control group. | 4, 8, 12 weeks
Change in QoL measured with QUALID from baseline to 12 weeks. Will be assessed in both the Intervention and Control group. | 12 weeks
Change in personal activity of daily living measured with the Physical Self Management Scale from baseline to 12 weeks. Will be assessed in both the Intervention and Control group. | 12 weeks
Nurses evaluation of systematic pain assessment tools by using a questionnaire developed for this study. Will be assessed in both the Intervention and Control group | 12 weeks
Pain management intervention applied when pain is detected with pain assessment tool Doloplus-2. Will be assessed for the Intervention group | 12 weeks
Validity and reliability of the Doloplus-2 pain scale. | 12 weeks
Convergent validity of three pain scales: the Doloplus-2, the Mobid-2 and the Checklist for non-verbal pain behavior. | Baseline - 12 weeks
Association between variables; pain, agitation, NPS, depression, ADL, QoL, analgesic use, psychotropic use Will be assessed in both the Intervention and Control group. | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liv Halvorsrud, PhD, Principal Investigator — Associate Professor
Locations (1):
- Faculty of Helath Science, Department of Nursing and Health Promotion, Oslo, PB 4 Saint Olavs Plass, Norway

IPD SHARING:
Plan to Share IPD: No